CLINICAL TRIAL: NCT06280781
Title: A Randomised Controlled Trial of Regular MRI Scans Compared to Standard Care in Patients With Prostate Cancer Managed Using Active Surveillance
Brief Title: Imperial Prostate 9 - ATLAS (Approaches To Long-Term Active Surveillance)
Acronym: IP9-ATLAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Queen Mary University of London (Other); University of Leeds (Other); University College, London (Other); University of York (Other); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 22CX7971; NIHR152027 (Other Grant/Funding Number: National Institute of Health Research - Health Technology Assessment)
Record Dates: First submitted 2024-01-25; First posted 2024-02-28 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Current (NICE defined active surveillance):
  PSA 3 monthly in year 1 and then 6 monthly with rectal exam annually. MRI will be carried out at 12 months (if not had one at diagnosis). A biopsy will be required if indicated due to changes in rectal exam or PSA.
  Planned (Regular MRI based active surveillance):
  Patients with a visible lesion or medium risk cancer will have PSA 6 monthly and MRI annually. All other patients will undergo PSA 6 monthly and MRI in years 1, 3 and 5. In all patients, a targeted biopsy will be carried out if the MRI PRECISE score is >/=4.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Control) Arm (No Intervention): PSA 3 monthly in year 1 and then 6 monthly with rectal exam annually. MRI will be carried out at 12 months (if not had one at diagnosis). If a diagnostic MRI was carried out, a 12 month MRI scan will not be required. A biopsy will be required if indicated due to changes in rectal exam or PSA. Follow-up for 5 years.
- Intervention Arm (Experimental): Patients with a visible lesion or medium risk cancer will have PSA 6 monthly and MRI scans annually. As per international PIRADS committee guidance the surveillance MRIs will be biparametric MRI scans which last approximately 15 minutes and exclude gadolinium contrast injection. All other patients will undergo PSA 6 monthly and MRI in years 1, 3 and 5. In all patients, a targeted biopsy will be carried out if the MRI PRECISE score is >/=4.
  Interventions: Diagnostic Test: MRI Scans

INTERVENTIONS:
Diagnostic Test: MRI Scans — The regular use of MRI in active surveillance will lead to greater confidence in active surveillance for patients with low and medium risk prostate cancer. This is because such a strategy is likely to detect cancer progression earlier with fewer invasive biopsies. Those patients randomised to the intervention arm will have additional MRI scans. These will be non-contrast so there is no risk from having repeated 1-2 yearly injections of gadolinium contrast. Patients with contraindications to MRI will not be taking part in the study so will not be exposed to an unnecessary MRI.
  Patients with a visible lesion or medium risk cancer will have PSA 6 monthly and MRI annually. All other patients will undergo PSA 6 monthly and MRI in years 1, 3 and 5. In all patients, a targeted biopsy will be carried out if the MRI PRECISE score is >/=4.
  Arms: Intervention Arm

SUMMARY:
The goal of this intervention study is for patients on active surveillance for prostate cancer, to demonstrate that use of regular MRI scans is better able to detect cancer progression over 5 years compared to the current NICE defined strategy.

Research Question P - In patients who are on active surveillance for low to medium risk prostate cancer, I - is the use of regular MRI scans C - compared to current NICE defined standard of care, O - better at detecting cancer progression with less cost to the NHS (fewer PSA tests, biopsies and clinic visits)?

Patients will be allocated in a 1.1 ratio to either MRI scans or the current NICE defined standard. Randomisation will be blocked (random block size) and stratified by MRI visibility of lesions (3 categories [ no visible lesion, diffuse changes, discrete visible lesion]), cancer Grade Group (GG1, GG2) and time since diagnosis. This study will not be blinded to patients or physicians.

DETAILED DESCRIPTION:
What is the problem being addressed?

Of 50,000 newly diagnosed patients with prostate cancer every year, about 7,600 choose active surveillance rather than immediate surgery or radiotherapy. Most have low risk whilst 20-30% have medium risk prostate cancer. This is because low and medium risk prostate cancers grow slowly. As a result, immediate treatment does not improve cancer-specific survival over 10 years but can cause high rates of urinary, sexual and bowel side-effects.

Although these cancers are slow growing, 25-34% will progress to higher risk over 5 years and need treatment later. Whilst there is no evidence that delayed detection of progression has an impact on survival, a recent systematic review has shown detrimental effects on other aspects of cancer control. For instance, in the largest RCT comparing active surveillance to immediate surgery or radiotherapy, 2-3 times as many patients had disease progression and cancer spread to other parts of the body in the active surveillance arm. So, active surveillance needs to be improved. NICE currently advise that active surveillance should involve 3-6 monthly prostate specific antigen (PSA) blood tests and rectal examinations. They advise an MRI and biopsy at 12 months. After one year, 3-6 monthly PSA and rectal examinations are recommended and further biopsy if the PSA starts to rise or if the rectal exam detects a prostate nodule.

This is problematic for 3 reasons:

First, PSA and rectal examination changes are inaccurate in detecting progression. As a result, some centres do regular biopsies every 1-2 years; this is borne out by a 48 physician survey (Jan 2022). However, biopsies alone are also inaccurate as they are ultrasound-guided; the operator can see the prostate but not areas suspicious for cancer progression.

Second, biopsies have side-effects such as infection, bleeding and pain; when these occur, patients are less likely to agree to further biopsies. Biopsies cost £488 and lead to significant NHS resource use. Regular and repeat biopsies can also cause prostate scarring making surgery more difficult if it is needed later.

Third, 10-43% of patients often decide to have treatment even if the cancer has not progressed. This is because of anxiety about living with cancer, or because of the biopsy and burden of tests. Some studies have shown other psychological impacts such as sub-clinical depression, illness uncertainty and hopelessness.

The Investigators propose using regular MRI scans in active surveillance to detect progression. The team led the pivotal UK studies which changed recommendations for MRI in diagnosing prostate cancer. Subsequently, The Investigators and others have shown that regular prostate MRI scans with targeted biopsies to areas of suspicion are accurate in ruling-out and detecting progression. To change NHS practice, an RCT is needed to compare regular MRI scans to current NICE defined standard of care in patients who choose active surveillance following an MRI-directed biopsy at time of diagnosis.

The studies proposal was positively reviewed by the NCRI Prostate Proposal Guidance panel (7/2/2022).

Why is this research important?

1. The regular use of MRI in active surveillance will lead to greater confidence in active surveillance for patients with low and medium risk prostate cancer. This is because such a strategy is likely to detect cancer progression earlier with fewer invasive biopsies. In previous studies, 1 of 672 patients chose treatment during surveillance due to anxiety.
2. An additional ~2000 patients with medium risk cancer could be managed with active surveillance in future.
3. Fewer NHS resources for clinic follow-ups, PSA tests and biopsies.

Of 5 research priorities that NICE have identified for prostate cancer, two relate to improving active surveillance. Similarly, the James Lind Alliance has 3 research priorities to improve active surveillance.

Research Question P - In patients who are on active surveillance for low to medium risk prostate cancer, I - is the use of regular MRI scans C - compared to current NICE defined standard of care, O - better at detecting cancer progression with less cost to the NHS (fewer PSA tests, biopsies and clinic visits)?

b) Aims and Objectives

Primary Objective

In patients on active surveillance for prostate cancer, to demonstrate that use of regular MRI scans is better able to detect cancer progression over 5 years compared to the current NICE defined strategy.

Difference between current and planned care pathways

Current (NICE defined active surveillance):

PSA 3 monthly in year 1 and then 6 monthly with rectal exam annually. MRI will be carried out at 12 months (if not had one at diagnosis). A biopsy will be required if indicated due to changes in rectal exam or PSA.

Planned (Regular MRI based active surveillance):

Patients with a visible lesion or medium risk cancer will have PSA 6 monthly and MRI annually. All other patients will undergo PSA 6 monthly and MRI in years 1, 3 and 5. In all patients, a targeted biopsy will be carried out if the MRI PRECISE score is >/=4.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above (no upper limit)
* Patients with a prostate (either cis-male gender or trans-female gender with no prior androgen deprivation hormone use at all).
* Diagnostic bi-parametric or multiparametric MRI
* Diagnostic systematic biopsy +/- targeted biopsy
* A histological diagnosis of localised prostate cancer
* Patient chosen active surveillance

Exclusion Criteria:

* On active surveillance for greater than 9 months prior to screening date.
* Contraindication to MRI or gadolinium contrast
* Previous hip replacement to both hips
* Contraindication to performing a biopsy guided by a transrectal ultrasound probe

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to disease type, prostate cancer is only found in male.
Enrollment: 1263 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Biopsy | 5 Years
  Progression in each group defined as higher risk cancer on biopsy (Grade Group >/=3)
  Prostate cancer progression rates and time to progression in each randomised arm defined on,
  • biopsy: grade progression to Grade Group 3 or greater or detection on biopsy of intraductal cancer or lymphovascular invasion. Many of our clinicians would include patients on active surveillance with cribriform pattern on Grade Group so this is not a factor for progression.
Staging | 5 Years
  Progression in each group defined as higher risk cancer on higher stage (>/=T3 or >/=N or >/=M1) over 5 years.
  Prostate cancer progression rates and time to progression in each randomised arm defined on,
  • staging: cancer has spread to surrounding tissues (extracapsular), lymph node involvement or distant body parts as demonstrated on cross-sectional imaging including MRI, CT, bone-scan or PET scans as deemed appropriate by the local multidisciplinary cancer team.

SECONDARY OUTCOMES:
Cost-effectiveness | 5 Years
  Cost-effectiveness of revising the prostate cancer active surveillance protocol to incorporate regular surveillance MRI within the NHS (QALYs questionnaire).
Biopsy Measurement | 5 years
  Biopsy would be recommended when there is a change on the MRI or if there is a consistent rise in PSA over 3 readings that is concerning for progression even if the MRI shows no change and other factors such as infection or prostatitis have been ruled out.
MRI & biopsy-related adverse events | 5 Years
  Patients will be asked to self-report pain and discomfort (referred to as pain hereafter) immediately after and seven days after biopsy on a 4-point Likert-type scale as none, mild, moderate, or severe. Specific related complications such as fever, flu-like shivers, pain, haematuria, haematochezia, and haemoejaculate will be self-reported at 35 to 90 days after prostate biopsy as absent or present following biopsy on a purpose designed questionnaire. For each symptom, patients will be asked to score the degree of "problem" as none, minor, moderate, or major. This will be used to derive a binary outcome for each symptom (present/moderate/severe problem vs. absent /minor problem).
Treatment | 5 Years
  Patients treatment options for progressive disease will be collected through multidisciplinary team (MDT) outcomes in the clinical records and clinic letters or entries by clinicians in the health records. Such options depending on cancer risk include; active surveillance, focal therapy, radical surgery or radiotherapy (with some men started on androgen deprivation therapy).
Compliance | 5 Years
  Compliance measured as proportion having each test (PSA, rectal exam, MRI) at each allocated timepoint and proportion agreeing to a biopsy when clinically recommended
EPIC Questionnaires | 5 years
  Annual changes in patient reported outcome measure (PROMS) using validated questionnaires, compared to baseline, to measure impact on urinary, erectile and bowel function (EPIC).
HADS Questionnaires | 5 Years
  Annual changes in patient reported outcome measure (PROMS) using validated questionnaires, compared to baseline, to measure impact on cancer-related anxiety (HADS)
EQ-5D-5L Questionnaires | 5 years
  Annual changes in patient reported outcome measure (PROMS) using validated questionnaires, compared to baseline, to measure impact on overall health-related quality of life (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Heatherwood Hospital, Ascot, Berkshire
  - Darent Valley Hospital, Dartford, Kent
  - Charing Cross Hospital, London

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT06280781/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT06280781/ICF_001.pdf